CLINICAL TRIAL: NCT06309264
Title: Benefits of Speech-based Audiometry and Low-gain Hearing Aids for Blast-exposed Veterans
Brief Title: Comparing Hearing Aid Fitting Methods in Blast-exposed Veterans
Acronym: SBA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Diego (Other); NADI Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: C5059-R; I01RX005059 (NIH)
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Auditory Diseases, Central
Keywords: blast injuries; occupational exposure; auditory diseases, central; hearing loss, hidden; hearing loss; hearing aids; hearing disorders; hearing loss, central; auditory perceptual disorders; correction of hearing impairment
MeSH Terms: conditions — Auditory Diseases, Central; Blast Injuries; Hearing Loss, Hidden; Hearing Loss; Hearing Disorders; Hearing Loss, Central; Auditory Perceptual Disorders

STUDY DESIGN:
Intervention Model Description: This study is a 2x2 randomized trial. Each subject receives a low-gain hearing aid. The randomized factors are:
  1. Fitting method. Half of the subjects have their hearing aids programmed using conventional methods based on the pure-tone audiogram. The remainder have their hearing aids programmed using the gain profile selected from speech-based audiometry.
  2. Daily hearing aid use. Half of the subjects will be assigned to use their hearing aids routinely in daily life for a six-week acclimatization period. The remaining half will be followed for the same six-week period but will use their hearing aids only to complete pre-post (mQuickSIN, fMRI) and weekly (DIN) laboratory assessments for speech recognition in noise. The daily use group will complete the same assessments.
  The factors are fully crossed such that there are four groups in the experiment.
Who Masked: Participant
Masking Description: Factor 1 is single blind: Participants will not know which procedure is used to program their hearing aid, but the investigator/outcomes assessor will. Factor 2 is unblinded: Participants will know whether they are assigned to the daily hearing aid use group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Speech-based hearing aid fitting (Experimental): Half of the study participants receive a hearing aid with gain settings determined via speech-based audiometry. Other hearing aid features such as noise reduction and directional microphones are disabled. Of this group of subjects, half are assigned to use the hearing aid daily for six weeks, while the remainder are followed for the same six-week period but use their hearing aids only to complete outcomes testing.
  Interventions: Device: Phonak Lumina P90
- Audiogram-based hearing aid fitting (Active Comparator): Half of the study participants receive a hearing aid with gain settings determined by applying the NAL-NL2 prescriptive formula to the pure-tone audiogram. Other hearing aid features such as noise reduction and directional microphones are disabled. Of this group of subjects, half are assigned to use the hearing aid daily for six weeks, while the remainder are followed for the same six-week period but use their hearing aids only to complete outcomes testing.
  Interventions: Device: Phonak Lumina P90

INTERVENTIONS:
Device: Phonak Lumina P90 — FDA approved hearing aid with gain settings determined either by speech-based audiometry or conventional fitting methods (NAL-NL2). Other features such as noise reduction and directional microphones are disabled for the duration of the study.

SUMMARY:
Since 2000, at least 250,000 U.S. Service members have experienced a blast-related mild traumatic brain injury. A retrospective analysis of over 100,000 post-9/11 Veterans shows that blast injury more than doubles the risk of a diagnosed auditory problem. Many blast-exposed Veterans experience "functional hearing difficulties" (FHDs): problems in challenging listening environments despite clinically normal hearing as measured by the pure-tone audiogram. VA audiologists have begun using low-gain hearing aids to treat FHDs, but there are no concrete guidelines for this application given standard procedures rely on the pure-tone audiogram. This study proposes a data-driven approach called speech-based audiometry (SBA), which optimizes hearing aid gains from a patient's responses to speech stimuli in aided conditions. This trial will assess the behavioral (speech recognition in noise, subjective listening difficulty) and neurophysiological (functional neuroimaging during a speech recognition task) benefits of low-gain hearing aids programmed conventionally or with SBA among blast-exposed Veterans with FHDs.

DETAILED DESCRIPTION:
The present study is a randomized trial of low-gain hearing aids in blast-exposed Veterans with normal or near-normal audiometric hearing and self-reported functional hearing difficulties. Hearing aids will be programmed using either conventional methods or a novel procedure called speech-based audiometry. Participants will be randomized into different groups receiving conventional or speech-based programming. Participants will be followed for a six-week intervention period and complete several outcome measures before, during, and after the intervention period. Each group will be further divided, at random, into equal subgroups assigned to (i) use their hearing aid daily during the six-week intervention period or (ii) use their hearing aid only to complete the outcomes assessments. The study will be broken into five periods:

1. Prescreening, screening, and enrollment
2. Preparatory period
3. Baseline
4. Treatment (first five weeks of hearing aid intervention)
5. Follow-up (final week of hearing aid intervention)

Prescreening, screening, enrollment (V0).

Prescreening includes identification of potential participants via medical record search, examination of patient rolls, clinician referral, or patient self-referral (e.g., from study advertisements). A prescreening phone call or in-person prescreening visit is scheduled for willing participants.

At the time of the in-person prescreening or prescreening phone call, a script will be used to learn if prospective participants meet basic eligibility criteria and are able to present for an in-person discussion of informed consent.

After prescreening is completed, potential participants meeting preliminary eligibility criteria will be scheduled for an initial study visit including informed consent procedures and, if consent is obtained, the following additional procedures.

Participants will be screened for inclusion and exclusion criteria. Screening includes performance of a routine audiological exam (otoscopy, tympanometry, air- and bone-conduction pure-tone audiometry) if a recent (< 6 months) exam is not available in the medical record. The subject also completes the following three questionnaires/interviews to determine eligibility, which are not part of routine audiological care:

1. Hearing Handicap Inventory for Adults (HHIA). The HHIA is a 25-item questionnaire that focuses on the emotional, social/situational, and occupational effects of hearing loss.
2. Mini-Mental State Exam (MMSE). The MMSE is an experimenter-led interview that assesses the global cognitive state of the subject including situational awareness, memory, language, and sensorimotor function.
3. Quantification of Cumulative Blast Exposure (QCuBE). The QCuBE is a semi-structured, experimenter-led interview that measures number and severity of exposures to blast, including date of exposure, distance from explosion, type of explosive, and protective gear worn, among other details. The QCuBE also obtains a brief history of non-blast head traumas.

   If a subject is not eligible (i.e. fails screening), an explanation is provided to the subject along with a full debriefing of the study. If a subject is eligible, they are randomized and asked to complete the following additional questionnaires:
4. Tinnitus Handicap Inventory (THI). The THI is a 25-item questionnaire that quantifies the impact of tinnitus on daily life.
5. Demographic data form (optional). This form obtains information on the subject's sex, ethnicity (Hispanic or Latino, not Hispanic or Latino), and race for reporting to the study sponsor using standard definitions.

Preparatory Period (V1, V2)

Two initial study visits will be conducted to prepare the subject for the hearing aid intervention. At the first visit (V1), the following procedures will be performed:

1. Speech-based audiometry. At the core of speech-based audiometry is the Open Speech Platform (OSP), an open-source hearing aid and speech processing platform with co-designed hardware and software elements. For the proposed work, the crucial component of OSP is a real-time master hearing aid, a modular software environment that abstracts the details of a digital hearing aid processor (e.g., block resampling, sub-band filtering, wide dynamic range compression, and feedback cancellation). That is, the master hearing aid is a software simulation of a hearing aid that performs all the same functions (e.g., sound amplification and compression). The flexible nature of the master hearing aid allows any arbitrary hearing aid prescription to be simulated in real time. The logic behind speech-based audiometry is as follows: (1) there is a library of potential hearing aid prescriptions (~1500 NAL-NL2 gain profiles) determined by unsupervised clustering performed on a large library of pure-tone audiograms from patients with a range of hearing loss levels and configurations; (2) there is also a library of speech stimuli (e.g., audiobook excerpts) that can be amplified with any prescription from the gain library in real time by OSP and presented to the patient over headphones; (3) this facilitates a non-exhaustive "search" of the possible prescriptions based on a patient's subjective ratings of speech amplified with different prescriptions; (4) in practice this takes the form of a series of A|B preference judgments made by the patient (much as in fitting for eyeglasses, "do you prefer A or B?"); (5) machine learning is used to select the A and B prescriptions for each presentation to optimize the search through the library of prescriptions for efficiency; (6) the procedure terminates when the search is finished.
2. Real ear measurement of realized gains. The real ear aided response (REAR) of the master hearing aid is obtained for the gain settings selected during speech-based audiometry following standard clinical procedures.
3. A hearing aid is ordered for the subject with preliminary gain settings established during speech-based audiometry or from the pure-tone audiogram (depending on group assignment).

At the second visit of the preparatory period (V2), real ear verification of hearing aid gain prescription is performed. That is, the preliminary gain settings initially programmed into the hearing aids are based on a set of "gain targets," which may differ from the actual gains realized when the hearing aids are worn by the subject. Thus, REAR measurements are again obtained for soft, moderate, and loud inputs separately for each ear. The hearing aid gains are manually adjusted by the fitting audiologist until the realized gains are within an acceptable range around the gain targets according to routine clinical standards. For subjects assigned to the speech-based audiometry group, the gain targets are the REAR measurements obtained during V1. For subjects assigned to the conventional fitting group, the gain targets are the output of the NAL-NL2 prescriptive formula applied to the subject's pure-tone audiogram; gains will be further adjusted based on the subject's subjective feedback, typically between 5-10 dB additional insertion gain at some or all frequencies between 500 and 4000 Hz. Once the final hearing aid gains are set, the hearing aids are placed in a hearing aid test box and their gain responses for soft, medium, and loud sounds are recorded. This will allow the study team to later use the hearing aid test box to verify that the hearing aid gains have not changed from prescribed settings. Finally, the subject will receive counseling from the fitting audiologist about how to use their hearing aids for the remainder of the study.

Baseline Period (V3, V4)

Study outcome measures will be obtained at baseline (i.e., before the daily use group has begun its six-week period of daily hearing aid usage). The first visit of the baseline period (V3) is an initial fMRI scan (see description of outcome measures). The fMRI scan session includes: (i) metal screening; (ii) counseling by a trained MRI technician about what to expect, how to remain safe, and how to trigger early termination of the MRI scan; (iii) a practice session conducted outside the scanner; (iv) familiarizing the subject with equipment to be used inside the scanner (e.g., button box, MR-compatible headphones) and placing the subject inside the MRI scanner; (v) acquisition of a T1 scout image and alignment of the MRI slices to be acquired in subsequent scans (axial slices aligned with the anterior-posterior commissure); (vi) acquisition of a high-resolution T1 anatomical scan and a gradient field mapping scan; (vii) eight fMRI scans; (viii) removal of the subject from the scanner; and (ix) 5-10 minute observation of the subject during a "cool off" period.

The second visit of the baseline period (V4) is a baseline speech-in-noise evaluation including the modified Quick Speech-In-Noise (mQuickSIN) test and the Digits in Noise (DIN) test in aided and unaided conditions. For subjects assigned to the daily hearing-aid-use group, hearing aids are dispensed to the subject for daily use over the next six weeks of the study.

Treatment Period (V5-V9)

Subjects complete weekly visits during the first five weeks of the six-week hearing aid intervention period (V5-V9). At each visit, the gain response of the subject's hearing aids will be verified in a hearing aid test box to ensure the final gain settings determined in V2 have not been altered. For subjects assigned to the daily hearing aid use group, the hearing aids' data loggers will also be checked to determine the number of hours the subject used the hearing aid each day since the preceding visit. The subject will complete the DIN as in V4.

Follow-Up Period (V10, V11)

At the end of the final week of the six-week hearing aid intervention period, subjects will complete two final visits (V10, V11) at which baseline testing is repeated. At V10, the subject completes a second fMRI scan with procedures just as in V3. At V11, the subject completes the same procedures as in V5-V9 with the following exceptions:

1. The subject also performs the mQuickSIN, as in V4.
2. The subject completes the THI, as in V0.
3. Subjects in the daily use group complete the Abbreviated Profile of Hearing Aid Benefit (APHAB). The APHAB is a validated questionnaire that measures subjective levels of listening difficulty pre and post hearing aid fitting in persons with hearing loss.

Once all the study procedures are completed, the subject receives a full debriefing. At the end of the debriefing, a study audiologist assumes the responsibility for transitioning the subject back to routine clinical care.

Instrumentation

Audiometric and speech-in-noise testing will be carried out in a double-walled sound-isolated audiometric chamber adjoined to a control room. Audiometric testing will be carried out using typical audiology equipment: A Madsen Astera2 or Grason-Stadler Audiostar Pro clinical audiometer calibrated to current standards (ANSI S3.6-2010) will be used to deliver the pure-tone signals for threshold testing through Etymotic Research ER-3A insert earphones. A Madsen Otoflex 100, Zodiac or Grasen-Stadler Tympstar Pro acoustic-immittance meter will be used for immittance measurements to verify normal middle ear function.

For speech-based audiometry, listeners will be seated comfortably in a sound-treated booth and wearing the same ER-3A earphones used in pure-tone audiometry. The procedure is driven by prototype commercial software (SpeechFit; Nadi, Inc.). Visual stimuli are displayed on a touchscreen monitor located in the sound booth. The same touchscreen monitor is used to collect responses from the subject. Acoustic stimuli are generated digitally by SpeechFit, output through a digital-to-analog converter and pre-amplifier (Motu M4), and amplified for presentation through ER-3A earphones. The equipment used for sound presentation is calibrated in Audcal software (Larson Davis, Inc.) to the same standard as routine speech recognition testing on a clinical audiometer (ANSI S3.6-2010). Calibration uses a Larson Davis 831C level meter and model AEC304 occluded ear simulator with calibrated 1/2-inch microphone.

An Auricle Freefit or Audioscan Verifit2 real ear measurement system connected to a VA-furnished and networked PC with installations of Otosuite and NOAH software will be used to collect real ear measurements. The same PC is used to program and order hearing aids.

For fMRI testing, speech stimuli will be presented over MR-compatible active noise cancelling headphones (Optoacoustics, Inc.). Amplification will be provided via the OSP master hearing aid running on the same PC used to generate and deliver the acoustic stimuli, with overall and band-specific levels verified by ear-canal probe microphone. In the aided condition, REAR will be matched as closely as possible to that recorded from the participant's fitted hearing aid. The MRI scanner is a 3 Tesla Siemens Skyra equipped with a 32-channel Siemens head coil, Philips SensaVue system for presentation of visual stimuli via MR-compatible LCD display, and Cedrus Lumina control box to collect button presses (Cedrus LS-LINE response box) and trigger signals from the scanner. Control of stimulus presentation is accomplished by custom MATLAB software running on a VA-owned PC that is permanently installed in the MRI control room.

The mQuickSIN is administered using software furnished by Walter Reed National Military Medical Center with sounds presented through a free field speaker array. The DIN is administered via custom Python software.

For all speech-in-noise tests (mQuickSIN, DIN, fMRI), unaided speech will be delivered at a moderate/conversational input level of 65 dB SPL.

ELIGIBILITY:
Inclusion Criteria:

Human subjects will be male or female Veterans selected without regard to race or ethnic background. All subjects will be 18 years of age or older and no more than 60 years old. On the QCuBE, all subjects must report at least one exposure to high-intensity blast (e.g., RPG, IED, mortar) close enough to feel the heat or pressure of the blast wave. All subjects must also score 20 or higher on the Hearing Handicap Inventory for Adults (HHIA). The remaining inclusion criteria for all subjects are:

1. pure-tone average (PTA) at 0.5, 1, 2, 4 kHz of 35 dB HL or better in each ear;
2. pure-tone thresholds no worse than 40 dB HL at any two audiometric frequencies up to 8 kHz;
3. no differences in pure-tone thresholds exceeding 10 dB between the two ears at more than one audiometric frequency up to 4 kHz;
4. native speaker of English; and
5. a score of at least 25 on the Mini Mental State Exam.

Exclusion Criteria:

1. a conductive hearing impairment or other otological pathology;
2. chronic disease or use of medication that might affect the auditory system or the subject's ability to perform the experimental tasks;
3. an inability to perform the experimental tasks;
4. any contraindications for MRI scanning (this may specifically exclude subjects who have a pacemaker, metal clips, or any other metal device in their body, or who have any other contraindication for MRI as determined by an MRI screening questionnaire); and
5. experience with hearing aids prior to the study.

Potential subjects meeting criterion 4 (contraindications for fMRI) will remain eligible to complete the non-MRI components of the trial (all visits other than V3, V10). These will be included in a Intent to Treat (ITT) cohort. Additional subjects who are eligible for MRI will be recruited into a Per Protocol (PP) cohort until the PP cohort meets target for total sample size (N = 60).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Quick Speech-in-Noise Test (mQuickSIN) Score at 6 weeks | Assessed at baseline (pre-intervention; V4) and at the end of the final week of the 6-week hearing aid intervention (V11). Results will be reported through study completion, on average once per year (aligned with the RPPR).
  Participants repeat back sentences embedded in four-talker babble, with each sentence presented at one of six signal-to-noise ratios decreasing from 33.5 dB to 8.5 dB in 5 dB steps. Each sentence is scored for number of correct keywords (out of five) and the total number correct over six sentences is subtracted by a normative value of 25.5 to obtain the "signal-to-noise ratio loss." The average signal-to-noise ratio loss across two sets of six sentences is obtained. The target sentences are time-compressed by 66% and subject to simulated room reverberation (0.25 s reverberation time). The outcome is the aided vs. unaided difference across all measurement time points (within-subject). The effect of hearing aid fitting method (conventional, speech-based) is obtained between-subjects. The effect of hearing aid acclimatization is the between-subject difference (daily use group vs. no daily use group) in the change of the aided vs. unaided difference at 6 weeks.
Abbreviated Profile of Hearing Aid Benefit (APHAB) | Assessed at the end of the final week of the 6-week hearing aid intervention (V11). Results will be reported through study completion, on average once per year (aligned with the RPPR).
  The APHAB is a validated questionnaire that measures subjective levels of listening difficulty pre and post hearing aid fitting in persons with hearing loss. The APHAB has been used to quantify subjective benefits of low-gain hearing aids in Service members with FHDs. The APHAB will be completed at the end of the study by participants assigned to use their hearing aids daily. The primary subjective study outcome is the aided vs. unaided difference in APHAB global score, obtained within-subject at a single time point (end of the final week of the six-week acclimatization period). The effect of hearing aid fitting method (conventional, speech-based) is obtained between-subjects.

SECONDARY OUTCOMES:
Change in Digits in Noise Test (DIN) Score at Weekly Intervals from Baseline to 6 weeks | Baseline (pre-intervention; V4), once per week during the hearing aid intervention period (V5, V6, V7, V8, V9), and once at the end of the final week of the 6-week hearing aid intervention (V11). Results will be reported through study completion, on aver
  Recordings of digit triplets (e.g., 5-3-8) are presented in a background of four-talker babble and the participant must enter the heard digits on a keypad. The background level is varied to target the signal-to-noise ratio (SNR) at which the target can be accurately recognized 50% of the time (SNR50). Target speech is subject to time compression (66%) and simulated reverberation (0.25 s). Two outcomes are obtained: the SNR50 and intraindividual variability in response times (RT-IIV) for SNR corresponding to 90% correct (estimated adaptively). The secondary outcome measures are thus the aided versus unaided difference, averaged across all measurement time points, in the SRT50 and RT-IIV (within-subject). The effect of hearing aid fitting method (conventional, speech-based) is obtained between-subjects. The effect of hearing aid acclimatization is the between-subject difference (daily use group vs. no daily use group) in the change of the aided vs. unaided difference at 6 weeks.

OTHER OUTCOMES:
Change in fMRI Activation at 6 weeks | Assessed at baseline (pre-intervention; V3) and at the end of the final week of the 6-week hearing aid intervention (V10). Results will be reported through study completion, on average once per year (aligned with the RPPR).
  Participants listen to sentences from the Coordinate Response Measure corpus. On each trial, a target sentence is spoken by a female talker and a competing sentence is spoken by a male talker (+3 dB target-to-masker ratio). The participant must identify keywords spoken by the talker from among three alternatives via button press. A total of 400 trials are performed with half amplified using the participant's fitted hearing aid gain settings (conventional or speech-based) and the remainder unamplified. The key outcome is the difference in activation (amplified vs. unamplified, within-subject) in a frontoparietal brain network defined in work conducted preliminary to the trial. The effect of hearing aid fitting method (conventional, speech-based) is obtained between-subjects. The effect of hearing aid acclimatization is the between-subject difference (daily use group vs. no daily use group) in the change of the amplified vs. unamplified contrast at 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Venezia, PhD, Principal Investigator — VA Loma Linda Healthcare System, Loma Linda, CA
Locations (3):
- United States (3):
  - VA Loma Linda Healthcare System, Loma Linda, CA, Loma Linda, California
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. Any IPD transmitted pursuant to a DUA will be coded using unique alphanumeric strings that are linked to the identity of individual subjects only in the master logbook stored at the primary site (VA Loma Linda Healthcare System).
  The Protocol, SAP, ICF, and CSR will be uploaded to clinicaltrials.gov following the Protocol Registration and Results System (PRS) procedures.
  Analytic code will be posted to the Open Science Framework under a unique study code registered to the PI (Dr. Venezia). This will include all code necessary to implement/collect the proposed outcome measures and to reproduce anonymous data elements (e.g., summary figures and tables) used in publications.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The Protocol, SAP, and ICF will be uploaded to clinicaltrials.gov prior to initiation of data collection. The CSR and Analytic Code will be uploaded within one year of the study end date.
  All of the above documents are expected to remain available for as long as the relevant web servers continue operating.
  LDS with IPD will become available within one year of the study end date and only upon request from a qualifying investigator or institution. The LDS will be available until destruction of identifiable data is mandated according to the VA Record Control Schedule.
Access Criteria: Sharing of LDS containing IPD requires full execution of a DUA between the VA Loma Linda Healthcare System and the requesting investigator/institution.